CLINICAL TRIAL: NCT02311881
Title: An Efficacy and Safety Study of Sustained-release Paracetamol in Subjects With Osteoarthritis
Brief Title: A 12-Week Efficacy Study of Paracetamol 1000mg Sustained-release Tablets in Patients With Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202195; RH02448 (Other: GSK)
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paracetamol 2000 mg twice daily (BID) (Experimental): Participants will be instructed to take two active paracetamol 1000 mg SR tablets twice daily (with 10-12 hours between adjacent doses) and two placebo to match paracetamol 665 mg SR tablets thrice daily (with 6-8 hours between adjacent doses) orally with approximately 8 ounces (~ 240 mL) of water/dose for 12 weeks.
  Interventions: Drug: Paracetamol 1000 mg SR tablets
- Paracetamol 1330 mg thrice daily (TID) (Active Comparator): Participants will be instructed to take two active paracetamol 665 mg SR tablets orally thrice daily (with 6-8 hours between adjacent doses) and two placebo to match paracetamol 1000 mg SR tablets orally twice daily (with 10-12 hours between adjacent doses) orally with approximately 8 ounces (~ 240 mL) of water/dose for 12 weeks.
  Interventions: Drug: Paracetamol 665 mg SR tablets
- Placebo (Placebo Comparator): Participants will be instructed to take two placebo to match paracetamol 1000 mg SR tablets twice daily (with 10-12 hours between adjacent doses) and two placebo to match paracetamol 665 mg SR tablets thrice daily (with 6-8 hours between adjacent doses) orally with approximately 8 ounces (~ 240 mL) of water/dose for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol 1000 mg SR tablets — Two paracetamol 1000 mg SR tablets administered orally two times a day plus two placebo-matched paracetamol 665 mg SR tablets administered orally three times a day for 12 weeks.
  Arms: Paracetamol 2000 mg twice daily (BID)
Drug: Paracetamol 665 mg SR tablets — Two paracetamol 665 mg SR tablets administered orally three times a day plus two placebo-matched paracetamol 1000 mg SR tablets administered orally two times a day for 12 weeks.
  Arms: Paracetamol 1330 mg thrice daily (TID)
Drug: Placebo — Two placebo-matched paracetamol 665 mg SR tablets administered orally three times a day plus two placebo-matched paracetamol 1000 mg SR tablets administered orally two times a day for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether paracetamol 1000 mg sustained-release (SR) tablets administered orally, twice daily are effective and safe in the treatment of patients with osteoarthritis of the knee or hip.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 40 and 80 years of age
* Diagnosis of moderate to moderately-severe osteoarthritis (OA) of either the knee or hip with respect to the following:

  * Pain in one knee/hip over 3 months immediately before screening visit
  * Use of non steroidal anti-inflammatory drugs (NSAIDs), acetaminophen (paracetamol) or any other analgesic for 3 or more days per week for at least 3 months prior to screening visit
  * Clinical diagnosis of osteoarthritis of knee/hip for minimum 6 month duration prior to screening visit
  * Therapeutic benefit with acetaminophen use with a score of ≥ 1 on 5-point categorical scale
  * Radiological evidence of ≥ Grade 2 osteoarthritis according to Kellgren-Lawrence radiographic criteria
* Increased WOMAC Pain Subscale score of at least 20 % following untreated run-in period
* Moderate to moderately-severe self-reported pain on a 5-point categorical scale following untreated run-in period
* Historical self-reported positive therapeutic benefit with paracetamol use for osteoarthritis pain relief

Exclusion Criteria:

* History of surgery or major trauma to the study joint
* Clinically significant signs or symptoms of inflammation upon completion of run-in period
* Required ongoing use of analgesic therapy for other indications, anticoagulants, psychotherapeutic agents, aspirin at daily doses greater than 325 mg, statin-class hypolipidemic agents at doses that have not been stabilized, or other treatments know to interfere with pain perception
* History of hepatic or renal or liver or biliary disease or gastrointestinal surgery
* Participants with alanine aminotransferase (ALT) >2 times Upper Limit Normal (2xULN) and bilirubin > 1.5 times Upper Limit Normal (1.5xULN) (However, if direct bilirubin is <35% and fractioned, isolated bilirubin >1.5xULN is acceptable)
* Other arthritis type, fibromyalgia or collagen vascular disease or secondary OA of study joint or chronic pain condition

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (49):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, North Hollywood, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Homestead, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Oldsmar, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evanston, Illinois
  - GSK Investigational Site, Prairie Village, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Watertown, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Hartsdale, New York
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Smithfield, Pennsylvania
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 57 centers in United States.
Pre-assignment Details: A total of 1531 participants were screened for study. Out of which only 960 participants who completed screening visit & took part in wash-out period were enrolled. Out of 960 enrolled participants, only 708 were randomized. 252 were not randomized because they did not fulfill specific inclusion criterion measured at the end of the wash-out period.
Groups:
- Paracetamol 2000 mg Twice Daily (BID): Participants were instructed to take two active paracetamol 1000 milligram (mg) sustained release (SR) tablets twice daily (with 10-12 hours between adjacent doses) and two placebo to match paracetamol 665 mg SR tablets thrice daily (with 6-8 hours between adjacent doses) orally with approximately 8 ounces ( ̴240 milliliter [mL]) of water/dose for 12 weeks.
- Paracetamol 1330 mg Thrice Daily (TID): Participants were instructed to take two active paracetamol 665 mg SR tablets orally thrice daily (with 6-8 hours between adjacent doses) and two placebo to match paracetamol 1000 mg SR tablets orally twice daily (with 10-12 hours between adjacent doses) orally with approximately 8 ounces ( ̴240 mL) of water/dose for 12 weeks.
- Placebo: Participants were instructed to take two placebo to match paracetamol 1000 mg SR tablets twice daily (with 10-12 hours between adjacent doses) and two placebo to match paracetamol 665 mg SR tablets thrice daily (with 6-8 hours between adjacent doses) orally with approximately 8 ounces ( ̴240 mL) of water/dose for 12 weeks.
Period: Overall Study
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Started | 235 (Started refers to all randomized participants.) | 236 (Started refers to all randomized participants.) | 237 (Started refers to all randomized participants.)
Safety Population | 234 (All treated participants: One participant was randomized but did not receive any treatment.) | 236 (All treated participants: One participant was randomized but did not receive any treatment.) | 237 (All treated participants: One participant was randomized but did not receive any treatment.)
Completed | 200 | 193 | 196
Not Completed | 35 | 43 | 41
Not completed — Did not meet the study criteria | 2 | 2 | 0
Not completed — Adverse Event | 7 | 15 | 8
Not completed — Lost to Follow-up | 3 | 3 | 2
Not completed — Protocol Violation | 1 | 2 | 3
Not completed — Withdrawal of consent | 14 | 16 | 17
Not completed — Other | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Subject has border line pregnancy test | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 4
Not completed — Sponsor Decision | 1 | 1 | 1
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Non-Compliance | 1 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Medical Monitor Discretion | 0 | 0 | 1
Not completed — Participant taking another medication | 0 | 0 | 1
Not completed — Serious Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are displayed for the safety population; i.e. for the population of all treated participants. One participant was randomized but did not receive any treatment.
Groups:
- Paracetamol 2000 mg Twice Daily (BID): Participants were instructed to take two active paracetamol 1000 mg SR tablets twice daily (with 10-12 hours between adjacent doses) and two placebo to match paracetamol 665 mg SR tablets thrice daily (with 6-8 hours between adjacent doses) orally with approximately 8 ounces ( ̴240 mL) of water/dose for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo | Total
Number analyzed (Participants) | 234 | 236 | 237 | 707
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.27 (8.544) | 60.47 (8.410) | 61.46 (8.187) | 60.73 (8.385)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 147 | 150 | 443
  Male | 88 | 89 | 87 | 264
Race/Ethnicity, Customized [Number; unit: number of participants]
  Hispanic or Latino | 77 | 81 | 95 | 253
  Not Hispanic or Latino | 157 | 155 | 142 | 454

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Mean Change From Baseline in Western Ontario McMaster (WOMAC) Pain Through Week 12 of Treatment
Description: The WOMAC Osteoarthritis Index is a 24-item questionnaire that assesses pain, physical function, and stiffness in the target joint. WOMAC Pain was measured using visual analogue scale (VAS) ranging from 0mm (no pain) to 100mm (extreme pain) at baseline and at week 1, 2, 4, 8, and 12. Lower values represent a better outcome. At each time point the assessment included 5 WOMAC Pain items: 1-walking on flat, 2-going up down stairs, 3-at night while in bed, 4-sitting or lying; 5-standing upright. Mean WOMAC Pain subscale score was calculated at each visit as the sum of 5 pain category scores divided by 5. Change from baseline was calculated for each visit as the mean WOMAC Pain subscale score minus the mean baseline WOMAC Pain subscale score. A negative change from Baseline indicated improvement. The time-weighted mean change was calculated as the area under the curve of change from baseline divided by the nominal time of the last on-therapy visit (week 12) from randomization (baseline).
Time Frame: Baseline up to week 12
Population: Modified intent to treat (mITT) population which included all participants included in the ITT population (included all randomized participants that received the study treatment & had at least one post-baseline efficacy assessment), except participants randomized in a site where good clinical practice issues were identified.
Measure: Least Squares Mean (Standard Error); unit: millimeter(mm)
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
millimeter(mm) | -28.25 (1.697) | -25.89 (1.714) | -25.74 (1.713)
Statistical Analysis 1: Comparison: Paracetamol 2000 mg Twice Daily (BID) vs Placebo; H0: There is no significant difference in mean change from baseline through week 12 of WOMAC Pain between twice daily Paracetamol 1000 mg SR tablets and placebo. H1: There is a significant difference in mean change from baseline through week 12 of WOMAC Pain between twice daily Paracetamol 1000 mg SR tablets and placebo; Test type: Superiority or Other; p = 0.1626, ANCOVA; LS mean difference = -2.51, 95% CI 2-sided [-6.037 to 1.016] — LS treatment means from mixed model analysis of covariance with treatment, target joint and center pools as fixed effects and baseline as a covariate
Statistical Analysis 2: Comparison: Paracetamol 2000 mg Twice Daily (BID) vs Paracetamol 1330 mg Thrice Daily (TID); H0: Difference in mean change from baseline through week 12 of WOMAC Pain between Paracetamol 1000 mg SR tablet and Paracetamol 665 mg SR tablet is ≤ - 5.3 (inferiority). H1: Difference in mean change from baseline through week 12 of WOMAC Pain between Paracetamol 1000 mg SR tablet and Paracetamol 665 mg SR tablet is > - 5.3 (noninferiority); Test type: Non-Inferiority or Equivalence — Paracetamol 2000mg BID is non-inferior to Paracetamol 1330mg TID if the upper bound of the 95% confidence Interval is less than 5.3; ANCOVA; LS mean difference = -2.36, 95% CI 2-sided [-5.894 to 1.166] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Paracetamol 1330 mg Thrice Daily (TID) vs Placebo; H0: There is no significant difference in mean change from baseline through week 12 of WOMAC Pain between Paracetamol 665 mg SR tablets and placebo. H1: There is a significant difference in mean change from baseline through week 12 of WOMAC Pain between Paracetamol 665 mg SR tablets and placebo; Test type: Superiority or Other; p = 0.9352, ANCOVA; LS mean difference = -0.15, 95% CI 2-sided [-3.687 to 3.394] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Time Weighted Mean Change From Baseline in WOMAC Physical Function Through Week 12 of Treatment
Description: The WOMAC Osteoarthritis Index is a 24-item questionnaire that assesses pain, physical function, and stiffness in the target joint. WOMAC Physical function was measured using VAS ranging from 0mm (no difficulty) to 100mm (extreme difficulty) at baseline and at week 1, 2, 4, 8, and 12. Lower values represent a better outcome. At each time point the assessment included 17 WOMAC Physical function categories. Mean WOMAC Physical function was calculated for baseline and each time point (sum of scores for 17 physical function categories divided by 17). Change from baseline was calculated for each visit as mean WOMAC physical function subscale score minus mean baseline WOMAC physical function subscale score. A negative change from Baseline indicated improvement. The time-weighted mean change was calculated as the area under the curve of change from baseline divided by the nominal time of the last on-therapy visit (week 12) from randomization (baseline).
Time Frame: Baseline up to Week 12
Population: Analysis for this outcome was conducted on mITT population which included all participants included in the ITT population (included all randomized participants that received the study treatment & had at least one post-baseline efficacy assessment), except participants randomized in a site where good clinical practices issues were identified.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
mm | -28.24 (21.341) | -26.23 (22.028) | -26.68 (20.137)

3. Secondary Outcome: Time Weighted Mean Change From Baseline in WOMAC Stiffness Through Week 12 of Treatment
Description: The WOMAC Osteoarthritis Index is a 24-item questionnaire that assesses pain, physical function, and stiffness in the target joint. WOMAC stiffness was measured using VAS ranging from 0mm (no stiffness) to 100mm (maximum stiffness) at baseline and at week 1, 2, 4, 8, and 12. Lower values represent a better outcome. At each time point the assessment included 2 WOMAC stiffness categories: 1- after awakening in the morning; 2- later in the day. Mean WOMAC stiffness was calculated for baseline and each time point (sum of scores for 2 stiffness categories divided by 2). Change from baseline was calculated for each visit as mean WOMAC stiffness subscale score at specific time point minus mean WOMAC stiffness subscale score at baseline. A negative change from Baseline indicated improvement. The time-weighted mean change from baseline was calculated as area under the curve of change from baseline divided by nominal time of the last on-therapy visit (week 12) from randomization (baseline).
Time Frame: Baseline up to week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
mm | -27.68 (21.579) | -25.61 (22.238) | -26.16 (21.554)

4. Secondary Outcome: Time-weighted Mean Change From Baseline in WOMAC Total Index Through Week 12 of Treatment
Description: The WOMAC Osteoarthritis Index is a 24-item questionnaire that assesses pain, physical function, and stiffness in the target joint. The Total Index Score included the WOMAC Pain Score (5 questions about pain where: 0=no pain to 100=extreme pain), the WOMAC Physical Function score (17 questions about the difficulty of daily activities where: 0=no difficulty to 100=extreme difficulty) and the WOMAC Stiffness Score (2 questions about stiffness where: 0=no stiffness to 100=extreme stiffness). WOMAC Total Index was calculated at baseline and each time point as sum of scores of all 24 WOMAC questions divided by 2400, ranging from 0 (no pain/difficulty/stiffness) to 1 (extreme pain/ difficulty/stiffness). Change from baseline was calculated as WOMAC Total Index at specific time point minus WOMAC Total Index at baseline. A negative change from Baseline indicated improvement.
Time Frame: Baseline up to week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
mm | -0.28 (0.209) | -0.26 (0.217) | -0.27 (0.200)

5. Secondary Outcome: Mean Change From Baseline in Global Patient Assessment of Arthritis (GPAOA)
Description: Participants performed an instantaneous GPAOA via a 0-100mm VAS, ranging from 0 (best ever) to 100 (worst ever) with respect to "With respect to your arthritis condition, how would you describe yourself now?" GPAOA was calculated periodically during the 12 week treatment period.
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: Analysis for this outcome was conducted on mITT population which included all participants included in the ITT population (included all randomized participants that received the study treatment & had at least one post-baseline efficacy assessment), except participants randomized in a site where good clinical practice issues were identified.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
mm
  At Baseline | 68.23 (16.965) | 69.20 (16.607) | 69.79 (16.734)
  At Week 4 | 39.34 (20.605) | 41.46 (22.330) | 42.93 (21.856)
  Change from baseline at Week 4 | -29.02 (22.343) | -27.78 (26.398) | -26.83 (24.229)
  At Week 8 | 36.08 (22.662) | 37.62 (23.523) | 39.09 (21.858)
  Change from baseline at Week 8 | -32.51 (24.429) | -31.15 (28.064) | -31.00 (23.649)
  At Week 12 | 32.41 (23.737) | 36.04 (23.848) | 35.44 (20.546)
  Change from baseline at Week 12 | -36.15 (26.192) | -33.04 (29.547) | -34.31 (25.521)

6. Secondary Outcome: Number of Participants Classified as Responder
Description: A participant was considered a "responder" if his/her improvement from baseline (change from baseline at week 12) satisfied at least one of the two criteria high' or 'moderate' improvement as follows:- High improvement: 50% improvement from baseline in the last available WOMAC pain score or 60% improvement from baseline in the last available WOMAC physical function score. Moderate improvement: Fulfills two out of three criteria: 30% improvement from baseline in the last available WOMAC Pain score, 20% improvement from baseline in the last available WOMAC Physical Function score, 25% improvement from baseline in the last available GPAOA.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Paracetamol 2000 mg Twice Daily (BID): Participants were instructed to take two active paracetamol 1000 mg SR tablets twice daily (with 10-12 hours between adjacent doses) and two placebo to match paracetamol 665 mg SR tablets thrice daily (with 6-8 hours between adjacent doses) orally with approximately 8 ounces (~ 240 mL) of water/dose for 12 weeks.
- Paracetamol 1330 mg Thrice Daily (TID): Participants were instructed to take two active paracetamol 665 mg SR tablets orally thrice daily (with 6-8 hours between adjacent doses) and two placebo to match paracetamol 1000 mg SR tablets orally twice daily (with 10-12 hours between adjacent doses) orally with approximately 8 ounces (~ 240 mL) of water/dose for 12 weeks.
- Placebo: Participants were instructed to take two placebo to match paracetamol 1000 mg SR tablets twice daily (with 10-12 hours between adjacent doses) and two placebo to match paracetamol 665 mg SR tablets thrice daily (with 6-8 hours between adjacent doses) orally with approximately 8 ounces (~ 240 mL) of water/dose for 12 weeks.
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
participants | 157 | 148 | 159

7. Secondary Outcome: Mean Change From Baseline in Daily Pain, Daily Stiffness and Pain/Stiffness (Composite) at Week 12
Description: Participants assessed their daily pain and stiffness each morning (upon awakening) during the 12-week treatment period using an 11-point Numerical Rating Scale (NRS), ranging from 0 (no pain / no stiffness) to 10 (extreme pain / extreme stiffness). Composite daily pain/stiffness score was calculated as sum of scores of pain and stiffness each morning divided by 2, ranging from 0 (no pain/stiffness) to 10 (extreme pain/stiffness). The mean of pain, mean of stiffness, and mean pain /stiffness composite score was calculated. Change from baseline was calculated as the difference between Daily Pain, stiffness and composite score each morning with that at baseline and was presented per week. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
score on a scale
  Pain at Baseline (n= 224, 225, 227) | 6.39 (1.902) | 6.27 (1.942) | 6.63 (1.774)
  Pain at Week 12(n= 176, 175, 177) | 3.80 (2.454) | 3.80 (2.197) | 3.82 (2.056)
  Pain, Change at Week 12 (n= 176, 175, 177) | -2.54 (2.301) | -2.49 (2.457) | -2.91 (2.442)
  Stiffness at Baseline (n= 224, 225, 227) | 6.20 (2.015) | 6.13 (1.908) | 6.38 (1.842)
  Stiffness at Week 12(n= 176, 175, 177) | 3.56 (2.383) | 3.63 (2.246) | 3.72 (2.145)
  Stiffness, Change at Week 12(n= 176, 175, 177 | -2.56 (2.227) | -2.44 (2.361) | -2.76 (2.500)
  Composite at Baseline (n= 224, 225, 227) | 6.30 (1.883) | 6.20 (1.817) | 6.51 (1.729)
  Composite at Week 12(n= 176, 175, 177) | 3.68 (2.361) | 3.71 (2.150) | 3.77 (2.043)
  Composite, Change at Week 12(n= 176, 175, 177 | -2.55 (2.209) | -2.46 (2.347) | -2.83 (2.410)

8. Secondary Outcome: Mean Number of Rescue Medication Pills Taken Per Day up to 12 Weeks
Description: Participants recorded use of rescue medication daily in their patient diary. The mean number of doses of rescue medications taken per day during the 12-week treatment period was calculated.
Time Frame: every day up to 12 weeks
Population: Analysis for this outcome was conducted on mITT population which included all participants included in the ITT population (included all randomized participants that received the study treatment & had at least one post-baseline efficacy assessment), except participant randomized in a site where good clinical practice issues were identified.
Measure: Mean (Standard Deviation); unit: number of rescue medication pills/day
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
number of rescue medication pills/day | 0.356 (1.7910) | 0.200 (0.8052) | 0.337 (1.1254)

9. Secondary Outcome: Mean Change From Baseline in Chronic Pain Sleep Inventory (CPSI)
Description: Chronic Pain Sleep Inventory (CPSI) was assessed, based on the three questions: CPSI-1-'Trouble falling asleep': How often the participant had trouble falling asleep? , CPSI-3-'Awakening due to pain at night': How often the subject was awakened by pain during the night, CPSI-4- Awakening due to pain in the morning': How often the participant was awakened by pain in the morning? The participants responded to these questions via 0-100mm VAS, ranging from 0 (never) to 100 (always). Sleep problem index (SPI) was calculated as mean of these three CPSI questions, ranging from 0 (never affected by pain during sleep) to 100 (always affected by pain during sleep).
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
mm
  At Baseline, CPSI-1 | 60.40 (26.089) | 57.77 (27.705) | 61.30 (25.500)
  At Baseline, CPSI-3 | 59.21 (26.980) | 57.19 (28.829) | 60.50 (25.532)
  At Baseline, CPSI-4 | 58.49 (27.759) | 56.94 (28.834) | 61.30 (25.773)
  At Baseline, Sleep Problems Index | 59.36 (25.886) | 57.26 (27.384) | 61.04 (24.156)
  At Week 4, CPSI-1 | 32.32 (25.396) | 29.23 (26.718) | 34.01 (24.701)
  At Week 4, Change in CPSI-1 | -27.87 (24.563) | -27.61 (28.248) | -27.44 (26.746)
  At Week 4, CPSI-3 | 32.54 (26.437) | 28.94 (27.232) | 32.75 (24.833)
  At Week 4, Change in CPSI-3 | -26.63 (25.621) | -27.51 (28.497) | -27.69 (26.257)
  At Week 4, CPSI-4 | 31.70 (25.667) | 28.85 (26.365) | 33.80 (25.749)
  At Week 4, Change in CPSI-4 | -26.55 (25.230) | -27.52 (28.135) | -27.47 (27.265)
  At Week 4, Sleep Problems Index | 32.16 (24.845) | 28.96 (26.102) | 33.52 (24.004)
  At Week 4, Change in Sleep Problems Index | -27.04 (23.458) | -27.59 (26.860) | -27.53 (24.930)
  At Week 8, CPSI-1 | 30.53 (26.672) | 29.22 (26.468) | 30.84 (24.277)
  At Week 8, Change in CPSI-1 | -29.98 (26.601) | -27.45 (28.842) | -31.34 (25.290)
  At Week 8, CPSI-3 | 30.25 (27.329) | 29.45 (27.286) | 29.71 (24.478)
  At Week 8, Change at CPSI-3 | -29.16 (27.321) | -26.91 (28.210) | -30.83 (25.892)
  At Week 8, CPSI-4 | 30.33 (26.856) | 29.12 (27.444) | 31.02 (24.625)
  At Week 8, Change at CPSI-4 | -28.19 (27.359) | -26.78 (29.961) | -30.11 (25.874)
  At Week 8, Sleep Problems Index | 30.33 (26.206) | 29.20 (26.533) | 30.50 (23.868)
  At Week 8, Change in Sleep Problems Index | -29.15 (25.838) | -27.11 (27.784) | -30.78 (24.315)
  At Week 12, CPSI-1 | 26.73 (25.302) | 26.90 (25.288) | 27.64 (21.977)
  At Week 12, Change in CPSI-1 | -33.12 (27.859) | -30.17 (30.532) | -34.43 (25.975)
  At Week 12, CPSI-3 | 26.95 (25.124) | 26.63 (25.684) | 27.42 (21.827)
  At Week 12, Change in CPSI-3 | -32.23 (29.228) | -29.99 (29.859) | -33.01 (27.116)
  At Week 12, CPSI-4 | 27.26 (25.887) | 26.85 (25.812) | 27.79 (22.581)
  At Week 12, Change in CPSI-4 | -30.90 (29.052) | -29.73 (30.967) | -32.97 (27.357)
  At Week 12, Sleep Problems Index | 26.96 (24.709) | 26.72 (25.135) | 27.61 (21.593)
  At Week 12, Change in Sleep Problems Index | -32.11 (27.489) | -30.03 (29.275) | -33.48 (25.485)

10. Secondary Outcome: Patient Global Assessment of Response to Therapy (PGART)
Description: The PGART is a global assessment of the participant's response to therapy, was measured using on a 5 point Likert scale as follows: 0=None (no good at all, ineffective), 1= Poor (some effect, but unsatisfactory), 2= Fair (reasonable effect, but could be better), 3= Good (satisfactory effect with occasional episodes of pain and/or stiffness), 4= Excellent (ideal response, virtually pain-free). Mean PGART scores from 5 point Likert scale was calculated periodically (at Week 4, Week 8, Week 12) for the 12 week treatment period.
Time Frame: Week 4, Week 8, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Number analyzed (Participants) | 224 | 225 | 227
score on a scale
  At Week 4 (n=197, 188, 202) | 2.50 (0.867) | 2.43 (0.871) | 2.25 (0.900)
  At Week 8(n=196, 184, 192) | 2.58 (0.852) | 2.40 (0.998) | 2.44 (0.958)
  At Week 12(n=189, 182, 181) | 2.62 (0.870) | 2.46 (1.022) | 2.43 (1.045)

ADVERSE EVENTS:
Time Frame: throughout the study completion (up to 408 days)
Arm/Group | Paracetamol 2000 mg Twice Daily (BID) | Paracetamol 1330 mg Thrice Daily (TID) | Placebo
Serious Adverse Events (participants affected / at risk) | 4/234 | 5/236 | 0/237
Other Adverse Events (participants affected / at risk) | 67/234 | 69/236 | 51/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paracetamol 2000 mg Twice Daily (BID) (N=234) | Paracetamol 1330 mg Thrice Daily (TID) (N=236) | Placebo (N=237)
CHEST PAIN (General disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 | 1 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paracetamol 2000 mg Twice Daily (BID) (N=234) | Paracetamol 1330 mg Thrice Daily (TID) (N=236) | Placebo (N=237)
NAUSEA (Gastrointestinal disorders) | 8 | 5 | 4
DIARRHOEA (Gastrointestinal disorders) | 6 | 7 | 2
FLATULENCE (Gastrointestinal disorders) | 4 | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 3 | 3 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 | 2 | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 2 | 1 | 1
VOMITING (Gastrointestinal disorders) | 2 | 2 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 6 | 2
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0 | 0
ODYNOPHAGIA (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 2 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 1 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 6 | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 3 | 2
BRONCHITIS (Infections and infestations) | 1 | 1 | 1
CONJUNCTIVITIS (Infections and infestations) | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 2 | 2
NASOPHARYNGITIS (Infections and infestations) | 1 | 3 | 2
SINUSITIS (Infections and infestations) | 1 | 1 | 4
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 1
FOLLICULITIS (Infections and infestations) | 0 | 1 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 2 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 2
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 5 | 5 | 5
DIZZINESS (Nervous system disorders) | 3 | 3 | 1
TENSION HEADACHE (Nervous system disorders) | 2 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 3 | 0 | 2
ASTHENIA (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 1 | 0 | 0
CHILLS (General disorders) | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 1 | 2
PERIPHERAL SWELLING (General disorders) | 1 | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7 | 4 | 0
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 | 0 | 0
BLOOD PRESSURE INCREASED (Investigations) | 0 | 1 | 1
HEPATIC ENZYME INCREASED (Investigations) | 0 | 3 | 0
HEPATITIS C VIRUS TEST POSITIVE (Investigations) | 0 | 0 | 1
LIVER FUNCTION TEST INCREASED (Investigations) | 0 | 1 | 0
LYMPHOCYTE COUNT INCREASED (Investigations) | 0 | 0 | 1
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 6 | 2 | 1
HOT FLUSH (Vascular disorders) | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 2 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 | 1 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 | 1 | 0
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
MILIARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0
URINE FLOW DECREASED (Renal and urinary disorders) | 1 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 2 | 1
RENAL PAIN (Renal and urinary disorders) | 0 | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0
URINE ODOUR ABNORMAL (Renal and urinary disorders) | 0 | 1 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 1 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1
DRY EYE (Eye disorders) | 1 | 0 | 0
RUBBER SENSITIVITY (Immune system disorders) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 1 | 1 | 0
RED BLOOD CELL ABNORMALITY (Blood and lymphatic system disorders) | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0
HYDROMETRA (Reproductive system and breast disorders) | 0 | 1 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 1 | 0
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.